CLINICAL TRIAL: NCT05455268
Title: Feasibility of e-Hematology Oncology Parents Education (eHOPE) for Information Support Among Malaysian Parents of Children With Hematological Cancer
Brief Title: Information Support Using an Online Learning Platform for Malaysian Pediatric Leukemia and Lymphoma Parents
Acronym: eHOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Collaborators: Universiti Putra Malaysia (Other); Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Tan Chai Eng, Principal Investigator, Universiti Kebangsaan Malaysia Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FF-2021-256; NMRR-21-613-58896 (Other: MREC Ministry of Health Malaysia)
Record Dates: First submitted 2022-06-27; First posted 2022-07-13 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Pediatric Acute Myeloid Leukemia; Pediatric Acute Lymphoid Leukemia; Pediatric Non-Hodgkin Lymphoma; Pediatric Hodgkin Lymphoma
Keywords: Information support; Online learning; Parent; Feasibility; Caregiver education; Self-efficacy; Knowledge
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Participants for both the intervention and control arms will be recruited simultaneously and allocated using block randomisation to achieve fairly equal numbers of participants in both study sites. At the end of the 8-week intervention period, participants in the waitlist control arm will receive access to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eHOPE (Experimental): Participants in the intervention group will receive access to e-Hematological Oncology Parent Education (eHOPE) and usual care. Participants will need to complete 4 self-paced activities over a period of 8 weeks. Each activity will be released at 2-weekly intervals.
  Interventions: Other: eHOPE; Other: Usual care
- Usual care (Active Comparator): Participants in the waitlist-control group will receive verbal explanations and caregiver education based on clinician's needs assessment in the course of their child's treatment process. At the end of 8-weeks, they will also receive access to eHOPE.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: eHOPE — e-Haematological Oncology Parents Education (eHOPE) consists of caregiving information for parents of children with leukaemia and lymphoma, presented in multimedia format through an online learning platform. The contents are developed in Malay language, encompassing basic information on disease and treatment, medical caregiving, emotional caregiving, appraising information, communication and self-care. Parents will be able to access multimedia information designed to support them in the care of their sick child. There are 4 self-paced activities in eHOPE with the following objectives:
  1. Parents should be able to outline key tasks related to care for their child at home.
  2. Parents should be able to outline strategies to initiate discussions with their child's healthcare providers.
  3. Parents should be able to appraise reliability of information sources.
  4. Parents should be able to identify coping strategies that they can use when faced with stressful situations.
  Arms: eHOPE
Other: Usual care — Face-to-face verbal discussions and caregiver training will be provided as deemed necessary by the clinicians.

SUMMARY:
This is a study protocol to determine whether it is feasible to support parents of children with blood cancers by providing information over an online learning platform. This study will be conducted in Malaysia. An online learning platform will be used to provide information relevant to parents who care for children diagnosed with leukemia or lymphoma. The use of this platform will be compared with current usual care, where only verbal discussions and ad hoc caregiver training is provided to support these parents, based on the clinician's judgement. Participants knowledge and confidence level in caregiving as well as coping will be compared between the two groups. To determine the feasibility of this method of information support, the researchers will also obtain feedback from participants who used the online learning platform and determine whether there are many who drop out from using it. The findings will determine whether use of online learning platform is suitable to deliver information support for parents, in view of currently limited resources for supportive care in childhood cancer care in Malaysia.

DETAILED DESCRIPTION:
This is the study protocol for a multi-centre interventional open-label randomized controlled feasibility trial to evaluate the feasibility of delivering informational support via an online learning platform to Malaysian parents of children with leukemia or lymphoma. The study will be conducted in two pediatric oncology centres in Kuala Lumpur, Malaysia. Study participants will include adult parents of children who were diagnosed with leukemia or lymphoma in the preceding 3. Block randomization will be used to allocate participants into the intervention or a waitlist-control arm. The intervention group will receive access to e-Hematological Oncology Parent Education (eHOPE), which provides information support for parents in the local Malay language, via an online learning platform. They will also receive usual care, which includes verbal explanations and caregiver education in the course of their child's treatment process. Parents will be able to access multimedia information designed to support them in the care of their sick child, and will need to complete 4 self-paced activities over a period of 8 weeks. The waitlist-control group will receive usual care, and at the end of 8 weeks, will also receive access to eHOPE. The primary outcome of this trial will be the change in caregiving knowledge, whereas secondary outcomes include caregiving self-efficacy and coping self-efficacy. Descriptive data on feasibility will include duration of recruitment to achieve targeted sample size, the drop-out rate of participants and identified barriers to implementation.

ELIGIBILITY:
Inclusion Criteria:

* Child (age <18 years) is diagnosed with either leukemia or lymphoma in the 3 months preceding recruitment
* Child is receiving care from either study site
* Able to access internet for health information via a computer, tablet or a mobile device
* Able to read and understand Malay language

Exclusion Criteria:

* Child is transferred to other hospital for continuation of treatment
* Extreme psychological distress
* Partner or spouse already enrolled into the current trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline caregiving knowledge at 8 weeks | At baseline and at 8 weeks
  This will be measured by the Hematological Oncology Parent's Education Caregiving Knowledge Questionnaire (HOPE-CKQ), a newly developed and validated 18-item Malay language questionnaire. The scale has a possible score range of 0-18. Higher scores will indicate better knowledge.
Recruitment rate | Through study completion, an average of 8 months
  This will be calculated as the number of participants recruited and randomized per centre per month.
Dropout rate | Through study completion, an average of 8 months
  This will be calculated as the proportion of participants who did not complete the trial over the total number of participants who were recruited and randomized.

SECONDARY OUTCOMES:
Change from baseline family caregiving self-efficacy at 8 weeks | At baseline and at 8 weeks.
  Based on scores of the Family Caregiving Activation in Transitions tool, a 10-item 6-point Likert scale with possible scores of 6 to 60. Higher scores indicate better caregiving self-efficacy.
Change from baseline coping self-efficacy at 8 weeks | At baseline and at 8 weeks.
  Based on scores of the Coping Self-Efficacy tool, a 26-item 11-point Likert scale with possible scores of 0 to 260. Higher scores denote better coping self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Chai Eng Tan, Principal Investigator — National University of Malaysia
Locations (2):
- Malaysia (2):
  - Hospital Tunku Azizah, Kuala Lumpur
  - Hospital Tunku Ampuan Besar Tuanku Aishah Rohani Hospital Pakar Kanak-kanak UKM (HPKK), Kuala Lumpur

IPD SHARING:
Plan to Share IPD: No
Due to requirements of the respective ethical committees, individual participant data will not be made available to other researchers. However, reasonable request for deidentified participant data may be considered by the principal investigator on case-to-case basis.

REFERENCES:
- [Background] Tan CE, Lau SCD, Latiff ZA, Lee CC, Teh KH, Sidik SM. Information needs of Malaysian parents of children with cancer: A qualitative study. Asia Pac J Oncol Nurs. 2021 Dec 25;9(3):143-152. doi: 10.1016/j.apjon.2021.11.001. eCollection 2022 Mar. PMID 35494095
- [Derived] Tan CE, Admodisastro N, Lau SCD, Tan KA, Teh KH, Lee CC, Mohd Sidik S. Development and user evaluation of an online caregiver education resource for Malaysian parents of children with leukemia or lymphoma. Asia Pac J Oncol Nurs. 2023 Dec 20;11(2):100363. doi: 10.1016/j.apjon.2023.100363. eCollection 2024 Feb. PMID 38304227

DOCUMENTS (1):
  • Informed Consent Form (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/68/NCT05455268/ICF_000.pdf